CLINICAL TRIAL: NCT03106389
Title: Misoprostol With And Without Transcervical Balloon Catheter In Second Trimester Termination Of Pregnancy: A Randomized Controlled Trial
Brief Title: Misoprostol With And Without Transcervical Balloon Catheter In Second Trimester Termination Of Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Alaa Elfeky, Professor of ObGyn, Ain Shams University, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBINTVN1
Record Dates: First submitted 2017-04-03; First posted 2017-04-10 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy Trimester, Second; Misoprostol; Catheters; Abortion, Second Trimester
Keywords: misoprostol; transcervical balloon catheter; second trimester; induced abortion
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: An open-label, parallel-arm, randomized controlled trial between two groups; each consisting of 54 women, undergoing termination of pregnancy during the second trimester for various medical reasons. The first group will receive 400 micrograms of misoprostol administered vaginally for the first dose, followed after 6 hours by 400 micrograms administered orally, repeated every 6 hours. The second group will receive the same regimen, but in addition will have a transcervical balloon (Foleys') catheter that will be inflated with 30 ml. of fluid; with weighted traction using a 1000 ml fluid-filled bag applying continuous pressure to the cervix. The target sample size is 108 cases randomized in a ratio of 1:1 using a computer-generated random sequence, allocation will be concealed in sealed, opaque consecutively-numbered envelopes. Women are counseled about the procedure, consenting women will be randomly assigned to one of the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol (Active Comparator): This group will receive 400 micrograms of misoprostol administered vaginally for the first dose, followed after 6 hours by 400 micrograms administered orally, repeated every 6 hours.
  Interventions: Drug: Misoprostol
- Misoprostol/Transcervical catheter (Experimental): This group will receive the same regimen, but will have in addition a transcervical balloon (Foleys') catheter that is inflated with 30 ml. of fluid; with weighted traction using a 1000 ml fluid-filled bag applying continuous pressure to the cervix
  Interventions: Drug: Misoprostol; Device: Misoprostol/Transcervical catheter

INTERVENTIONS:
Drug: Misoprostol — 400 micro grams misoprostol administered vaginally followed every 6 hours by 400 micro grams orally until complete expulsion
  Other Names: Cytotec; Misotac
Device: Misoprostol/Transcervical catheter — Foleys' catheter introduced into the cervix and inflated with 30 ml. of fluid; weighted traction applied by using a 1000 ml fluid-filled bag
  Other Names: Foley catheter
  Arms: Misoprostol/Transcervical catheter

SUMMARY:
This randomized controlled study will be performed to compare the benefits and risks associated with the administration of misoprostol with or without the use of a transcervical balloon catheter to terminate pregnancy in the second trimester (defined as gestational age between 14 and 28 weeks of gestation).

DETAILED DESCRIPTION:
The study will be conducted at Ain Shams Maternity Hospital. An open-label, parallel-arm, randomized controlled trial between two groups; each consisting of 54 women, undergoing termination of pregnancy during the second trimester for various medical reasons. The first group will receive the standard misoprostol protocol for termination of second trimester pregnancy currently practiced at Ain Shams Maternity Hospital; 400 micrograms of misoprostol administered vaginally for the first dose, followed after 6 hours by 400 micrograms administered orally, repeated every 6 hours till complete expulsion of the uterine contents or surgical interference is decided. The second group will receive the exact same regimen, but will have in addition a transcervical balloon (Foleys') catheter that will be inflated with 30 ml. of fluid; and will have weighted traction applied to the catheter through using a 1000 ml fluid-filled bag in order to apply continuous pressure to the cervix. The target sample size was calculated to be 108 cases; randomization will be in a ratio of 1:1 using a computer-generated random sequence. Allocation will be concealed using sealed, opaque consecutively-numbered envelopes. Women are counseled about the procedure, consenting women will thus be randomly assigned to one of the groups.

ELIGIBILITY:
Inclusion Criteria: pregnancy in the second trimester (defined as gestational age between 14 and 28 weeks of gestation) with a medical indication for termination of pregnancy.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 108 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-07-31 (Estimated)

PRIMARY OUTCOMES:
Induction-expulsion interval | 48 hours from starting intervention
  The duration from the administration of the first misoprostol dose vaginally till complete expulsion of the uterine contents; complete uterine emptiness will be confirmed by ultrasonographic assessment

SECONDARY OUTCOMES:
Total required doses of misoprostol | 48 hours from starting induction
  The total amount of misoprostol used per participant during the procedure
The need for surgical interventions | 1 week from starting induction
  The number of participants requiring any surgical intervention under anesthesia to complete uterine emptiness

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Elfeky, Professor, Principal Investigator — AinShams University Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo Governorate, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after publication of the study upon formal request by researchers and research centers that collaborate with Ain Shams Maternity Hospital. Data could be obtained through contacting PI by email.